CLINICAL TRIAL: NCT03318003
Title: Auto-PAP Therapy For Improved Fetal Growth
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: ResMed Foundation (Other)
Responsible Party: Principal Investigator, Louise O'Brien, Associate Professor, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HUM00132040; N023548 (Other Grant/Funding Number: ResMed Foundation)
Record Dates: First submitted 2017-10-13; First posted 2017-10-23 (Actual); Results first posted 2022-01-25 (Actual); Last update posted 2022-11-18 (Actual); Status verified 2022-11

CONDITIONS: Obstructive Sleep Apnea; Pregnancy
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Auto-PAP Therapy (Experimental)
  Interventions: Device: Auto-PAP
- No Therapy (No Intervention)

INTERVENTIONS:
Device: Auto-PAP — Women will be using the Auto-PAP device nightly from randomization to end of pregnancy
  Arms: Auto-PAP Therapy

SUMMARY:
The purpose of this study is to see whether the presence of night-time breathing disturbances ("sleep-disordered breathing") in pregnant women is related to fetal growth patterns. The hypothesis is that fetal growth slows in the 3rd trimester in women with sleep-disordered breathing. Use of a nighttime breathing therapy called auto-PAP could minimize the slowing in fetal growth.

ELIGIBILITY:
Inclusion Criteria:

* at least 18 years old;
* no more than 20 weeks pregnant;
* pregnant with one baby;
* found to have sleep-disordered breathing as measured by a sleep study. If you are found to have severe sleep apnea on the sleep study you will be referred for clinical care instead of participating in the study.

Exclusion Criteria:

* more than 20 weeks pregnant;
* pregnant with twins, triplets, or more babies;
* a current smoker, drink alcohol, or use recreational drugs;
* currently using positive-airway pressure therapy for treatment of obstructive sleep apnea;
* diagnosed with certain conditions such as bullous lung disease, a bypassed upper airway, pneumothorax (collapsed lung), pneumocephalus (leak of cerebrospinal fluid, the fluid that the brain and spine float in), if you have had recent trauma, or recent nasal surgery.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2017-12-01 (Actual); Primary Completion 2020-08-03 (Actual); Study Completion 2020-08-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Louise M O'Brien, PhD, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan Heath System, Ann Arbor, Michigan, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- No Therapy: No treatment
Period: Overall Study
Arm/Group | Auto-PAP Therapy | No Therapy
Started | 21 | 22
Completed | 20 (completed means the presence of 3rd trimester ultrasound and delivery information.) | 20
Not Completed | 1 | 2
Not completed — Withdrawal by Subject | 1 | 1
Not completed — fetal loss | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Auto-PAP Therapy | No Therapy | Total
Number analyzed (Participants) | 21 | 22 | 43
Age, Continuous [Mean (Standard Deviation); unit: years] | 29.7 (4.4) | 34.4 (4.2) | 32.2 (4.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 22 | 43
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 2 | 3
  Not Hispanic or Latino | 20 | 20 | 40
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 7 | 1 | 8
  White | 14 | 20 | 34
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 21 | 22 | 43
gestational age at enrollment [Mean (Standard Deviation); unit: weeks] | 17.1 (4.4) | 17.2 (4.1) | 17.1 (4.2)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Slowing of Fetal Growth by 33% or More During the Last Trimester
Description: A slowing of fetal growth will be defined as a slowing of fetal growth by >=33% during the last trimester
Time Frame: 3rd trimester
Population: Because the latter part of the study was overlapping March 2020, some women did not get all of their research ultrasounds. Data below is shared for all women for whom at least one 3rd trimester ultrasound is available.
Measure: Count of Participants; unit: Participants
Arm/Group | Auto-PAP Therapy | No Therapy
Number analyzed (Participants) | 18 | 21
Participants | 8 | 8
Statistical Analysis 1: Comparison: Auto-PAP Therapy vs No Therapy; Test type: Superiority; p = 0.92, Chi-squared — no adjustments made; Pearson Chi Square = 0.76

2. Secondary Outcome: Presence or Absence of Placental Hypoxia
Description: The placenta will be reviewed by a pathologist to determine the presence or absence of areas of hypoxia
Time Frame: At delivery the placenta will be collected and processed.
Population: Some placentas were not collected and sent to pathology as intended, perhaps in part because of fewer staff available during the COVID inflected months.
Measure: Count of Participants; unit: Participants
Arm/Group | Auto-PAP Therapy | No Therapy
Number analyzed (Participants) | 13 | 15
Participants
  Hypoxia determinations | 1 | 4
  Non-hypoxia determinations | 12 | 11

ADVERSE EVENTS:
Time Frame: through delivery up to a maximum of 33 weeks
Arm/Group | Auto-PAP Therapy | No Therapy
All-Cause Mortality (participants affected / at risk) | 0/21 | 0/22
Serious Adverse Events (participants affected / at risk) | 0/21 | 2/22
Other Adverse Events (participants affected / at risk) | 0/21 | 0/22
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Auto-PAP Therapy (N=21) | No Therapy (N=22)
Demise (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 2 (2) — Fetal/infant demise

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-04-10): https://cdn.clinicaltrials.gov/large-docs/03/NCT03318003/Prot_SAP_000.pdf